CLINICAL TRIAL: NCT05470959
Title: Bioactive Ionic Resin Composite Versus Resin-Modified Glass Ionomer Cavity Liners: 2-Year Randomized Clinical Trial
Brief Title: Bioactive Composite Versus Resin-Modified Glass Ionomer Liners: 2-Year Clinical Trial
Acronym: BIRCRMGILYCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M19091019
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACTIVA bioactive (Other): bioactive ionic resin composite
  Interventions: Other: ACTIVA bioactive
- Riva LC (Other): Resin-modifed glass ionomer
  Interventions: Other: Riva LC

INTERVENTIONS:
Other: ACTIVA bioactive — bioactive ionic resin composite
  Arms: ACTIVA bioactive
Other: Riva LC — resin-modified glass ionomer
  Other Names: Riva light cure
  Arms: Riva LC

SUMMARY:
compare 2-year clinical performance of recent bioactive ionic resin composite to resin-modified glass ionomer liner in indirect dental pulp treatment.

DETAILED DESCRIPTION:
patients were enrolled in the clinical trial. Each patient had two deep carious lesions, one on each side of the mouth. After selective caries removal, cavities were lined with bioactive ionic resin composite (Activa Bioactive Liner/Base) or resin-modified glass ionomer liner (Riva Light Cure RMGI). All cavities were then restored with nanofilled resin composite (Filtek Z350xt). All materials were placed according to the manufacturers' instructions. Clinical evaluation was accomplished using World Dental Federation (FDI) criteria at baseline and after 6 months, one year, one and half years, and two years.

ELIGIBILITY:
Inclusion Criteria:

* presence of two deep carious lesions, one on each side of the mouth (ICDAS 5 or 6)
* vital teeth
* no sensitivity to teeth percussion
* no spontaneous pain
* no radiolucency in the periapical or furcation area of teeth
* complete and normal occlusion
* good oral hygiene

Exclusion Criteria:

* poor oral hygiene
* severe or chronic periodontal problems
* periapical lesions
* heavy bruxism
* non-vital teeth
* visibly cracked teeth
* spontaneous dental pain
* sensitivity to teeth percussion

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
assess clinical performance of bioactive ionic resin composite and resin-modified glass ionomer liner by using FDI clinical criteria | 2-years
  comparison of 2-year clinical performance of recent bioactive ionic resin composite( ACTIVA bioactive) to resin-modified glass ionomer liner ( Riva LC) in indirect dental pulp treatment using FDI world dental federation clinical criteria.

CONTACTS AND LOCATIONS:
Overall Officials: salah mahmoud, professor, Study Director — faculty of dentistry, mansoura university
Locations (1):
- Faculty of Dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed B, Wafaie RA, Hamama HH, Mahmoud SH. 3-year randomized clinical trial to evaluate the performance of posterior composite restorations lined with ion-releasing materials. Sci Rep. 2024 Feb 28;14(1):4942. doi: 10.1038/s41598-024-55329-6. PMID 38418863